CLINICAL TRIAL: NCT01612702
Title: The Use of a Single, Low-dose Dexamethasone in Total Knee Arthroplasty
Brief Title: Efficacy and Safety of Single, Low-dose Dexamethasone in Patients After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tae Kyun Kim (Other)
Responsible Party: Sponsor-Investigator, Tae Kyun Kim, Direcor, Joint reconstruction center, SNUBH, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1102/121-006
Record Dates: First submitted 2012-06-03; First posted 2012-06-06 (Estimated); Results first posted 2013-05-21 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Osteoarthritis, Knee
Keywords: postoperative nausea and vomiting; postoperative pain
MeSH Terms: conditions — Osteoarthritis, Knee; Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Experimental): dexamethasone 10 mg administration 1 hour before surgery
  Interventions: Drug: Dexamethasone
- Control (No Intervention): No dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 10 mg intravenous administration
  Arms: Dexamethasone

SUMMARY:
This study was conducted to determine the efficacy of an additional preemptive, single, low-dose dexamethasone in terms of incidence and severity of postoperative nausea/vomiting (PONV), pain level, and the safety in terms of wound complications in patients managed with our antiemetic protocol based on Ramosetron following TKA.

DETAILED DESCRIPTION:
Postoperative pain and emesis can cause postoperative systemic complications and delay recovery and rehabilitation in patients following total knee arthroplasty (TKA). Furthermore, patients who suffered from severe postoperative pain and emesis tend to be dissatisfied with their surgical treatments. Although contemporary protocols to control perioperative pain and emesis after TKA have been reported to substantially reduce postoperative pain and emesis compared with traditional measures, pain and emesis after TKA remain to be a challenging issue for patients and health care providers. In our previous study, the use of Ramosetron was found to reduce postoperative emetic events, but the antiemetic effects by Ramosetron were incomplete. In search of a further antiemetic measure, we identified the use of dexamethasone as the additional measure fortifying our antiemetic protocol using Ramosetron.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary osteoarthritis, knee
* Scheduled for elective total knee arthroplasty
* Signed written informed consent

Exclusion Criteria:

* Refusing participate
* Contraindication to regional anesthesia
* Severe impairment of bowel motility
* administration of other antiemetic drug within 24hours before surgery
* systemic steroid within 24hours before surgery
* history of cardiovascular & respiratory disease
* renal & hepatic failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T K Kim, MD, PhD, Principal Investigator — Joint Recontruction Center, Seoul National University Bundang hospital
Locations (1):
- Joint Reconstruction Center, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 305 patients who were scheduled for unilateral total knee arthroplasty at Seoul National Bundang Hospital from April 2011 to December 2011 were recruited.
Pre-assignment Details: 14 patients were excluded before assignment. 5 were other diagnosis such as rheumatoid arthritis, secondary osteoarthritis, 4 had serious medical conditions such as renal failure, heary failure, 5 refused to participate
Period: Overall Study
Arm/Group | Dexamethasone | Control
Started | 146 | 145
Completed | 135 | 134
Not Completed | 11 | 11
Not completed — Protocol Violation | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Control | Total
Number analyzed (Participants) | 146 | 145 | 291
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 132 | 131 | 263
Age Continuous [Mean (Standard Deviation); unit: years] | 72 (6.7) | 72 (6.2) | 72 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 119 | 236
  Male | 29 | 26 | 55
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 146 | 145 | 291

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Nausea and Vomiting
Description: A clinical investigator who is blinded to randomization assessed the incidence of postoperative nausea which defined as subjective unpleasant sensation associated with awareness of the urge to vomit and as emetic episode and vomiting
Time Frame: within 72 hours after surgery
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Dexamethasone | Control
Number analyzed (Participants) | 146 | 145
percentage of participant | 24 [22.8 to 25.2] | 40 [38 to 42]

2. Secondary Outcome: Pain Level
Description: A blinded investigator asked participants to recall the most severe pain level during 6 to 24 hour after surgery using with a visual analogue scale that ranged from 0 (no pain) to 10 (worst imaginable pain).
Time Frame: 6 to 24 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexamethasone | Control
Number analyzed (Participants) | 146 | 145
units on a scale | 2.4 (1.0) | 4.0 (2.0)

3. Secondary Outcome: Wound Complication
Description: Number of participants with a sinus tract communicating with the prosthesis; a pathogen was isolated by culture from tissue or fluid samples taken from the affected joint; tests revealed elevated serum erythrocyte sedimentation rate (ESR) or serum C-reactive protein (CRP) concentration with elevated synovial white blood cell (WBC) count or neutrophil percentage; or pus discharge from the affected joint was present within 30 days after total knee arthroplasty were measured.
Time Frame: within 30 days after surgery
Measure: Number; unit: participant
Arm/Group | Dexamethasone | Control
Number analyzed (Participants) | 146 | 145
participant | 1 | 1

ADVERSE EVENTS:
Time Frame: 30 days after total knee arthroplasty
Description: wound complication such as postoperative infection, wound dehescence.
Arm/Group | Dexamethasone | Control
Serious Adverse Events (participants affected / at risk) | 1/146 | 1/145
Other Adverse Events (participants affected / at risk) | 0/146 | 0/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=146) | Control (N=145)
Wound complication (Surgical and medical procedures) | 1 (1) | 1 (1) — wound compltications within 30 days after total knee arthroplasty

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes